CLINICAL TRIAL: NCT04559048
Title: Investigation of Pain Incidence After FK506 Immunosuppressive Therapy in Liver Transplantation Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HBTS1411206
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Liver Transplantation
Keywords: Chronic Pain; Liver Transplantation; FK506
MeSH Terms: conditions — Chronic Pain | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FK506-treated group: In FK506-treated group, the patients who underwent liver transplant are treated with FK506 immunosuppressive therapy.
  Interventions: Drug: FK506
- control group without FK506 treatment: In control group, the patients who underwent liver transplant are treated without FK506.

INTERVENTIONS:
Drug: FK506 — FK506 (tacrolimus), a calcineurin inhibitor, is widely used as an immunosuppressant to lower the risk of organ rejection after organ transplantation
  Groups: FK506-treated group

SUMMARY:
FK506 (tacrolimus), a calcineurin inhibitor, is widely used as an immunosuppressant to lower the risk of organ rejection after organ transplantation, and to treat T cell-mediated diseases such as eczema and atopic dermatitis. FK506 treatment often accompanies pain sensation in patients with atopic dermatitis or after organ transplantation. In previous studies, the investigators confirmed that FK506 treatment increased neuronal activity of primary afferent neurons and causes pain behavior in naïve mice. In order to further search for objective clinical evidence, the investigators proposed to investigate pain incidence after FK506 immunosuppressive therapy in liver transplantation patients. The investigators will investigate pain incidence and pain intensity in patients who underwent liver transplant from September of 2011 to May of 2018 in the Liver Health Rehabilitation Association. The patients who were divided into two groups based on whether or not FK506 was used in the immunosuppressive therapy. The patients in control group (without FK506 treatment) and FK506-treated group report pain sensation 3 months and 12 months after liver transplant. The investigators will compare the pain incidence between the two groups at both time points. On the other hand, the investigators will further investigate changes in pain sensation after 1st and 2nd reductions of FK506 dose. Pain is reported subjectively by the patient using the visual analogue scale (VAS) 1 month after dose reduction. In our study, 1st and 2nd reductions of FK506 dose refers to the first two dose-adjustments (approximately 6 months apart) that occurred 3-6 months after the liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. had liver transplantation for end-stage liver disease
2. was ≥18 years of age at the time of liver transplantation -

Exclusion Criteria:

1. liver cancer
2. acute (fulminant) liver failure
3. multiorgan transplant
4. chronic postsurgical pain
5. fibromyalgia, osteoarthritis, low back pain and inflammatory pain of any origin
6. peripheral and central neuropathic pain of any origin
7. chronic secondary visceral pain
8. chronic cancer-related pain that is due to cancer or its treatment -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A retrospective study was conducted in patients who underwent liver transplant from September of 2011 to May of 2018 in the Liver Health Rehabilitation Association(China)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
pain incidence | within 2 years after liver transplantation
  Pain is defined as painful sensation that lasts or recurs for 1-3 months within 3 months after liver transplantation, or for longer than 3 months within 12 months after liver transplantation.
pain intensity | within 2 years after liver transplantation
  Pain is reported subjectively by the patient using the visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Dequn Liu, M.D., Study Chair — The Second Hospital of Tangshan
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Background] Reitamo S, Rustin M, Ruzicka T, Cambazard F, Kalimo K, Friedmann PS, Schoepf E, Lahfa M, Diepgen TL, Judodihardjo H, Wollenberg A, Berth-Jones J, Bieber T; European Tacrolimus Ointment Study Group. Efficacy and safety of tacrolimus ointment compared with that of hydrocortisone butyrate ointment in adult patients with atopic dermatitis. J Allergy Clin Immunol. 2002 Mar;109(3):547-55. doi: 10.1067/mai.2002.121832. PMID 11898005
- [Background] Malat GE, Dupuis RE, Kassman B, Rhoads JM, Freeman K, Lichtman S, Johnson MW, Gerber D, Andreoni K, Fair J. Tacrolimus-induced pain syndrome in a pediatric orthotopic liver transplant patient. Pediatr Transplant. 2002 Oct;6(5):435-8. doi: 10.1034/j.1399-3046.2002.02030.x. PMID 12390434